CLINICAL TRIAL: NCT02182869
Title: Safety Assessment of Cumulative Dose of Combivent® HFA-propelled Metered Dose Inhaler in Comparison to Combivent® CFC-propelled Metered Dose Inhaler. A Randomised, Double-blind, Active-controlled, Two-way Cross-over Study in COPD Patients
Brief Title: Combivent® HFA-propelled Compared to CFC-propelled Metered Dose Inhaler in Patients With COPD (Chronic Obstructive Pulmonary Disease)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1012.43
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (2):
- Combivent® HFA (Experimental)
  Interventions: Drug: Combivent® HFA inhalation aerosol
- Combivent® CFC (Active Comparator)
  Interventions: Drug: Combivent® CFC inhalation aerosol

INTERVENTIONS:
Drug: Combivent® HFA inhalation aerosol
  Arms: Combivent® HFA
Drug: Combivent® CFC inhalation aerosol
  Arms: Combivent® CFC

SUMMARY:
Study to evaluate the safety of combivent delivered in two different formulations (hydrofluoroalkane (HFA) or chlorofluorocarbon (CFC)) from a metered dose inhaler (MDI), using a cumulative dose response model in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 40 years of age or older
2. A diagnosis of COPD as defined by American Thoracic Society (ATS) criteria. Patients must have relatively stable, moderate to severe airway obstruction with a baseline FEV 1 <=65% of predicted normal and FEV1/FVC >=70%.
3. A smoking history of more than ten pack-years. A pack-year is defined as the equivalent of smoking one pack of 20 cigarettes per day for a year
4. Able to perform technical satisfactory pulmonary function test
5. Able to be trained in the proper use of a MDI
6. Having signed an informed consent from prior to participation in the trial
7. Affiliation to the French social security system or beneficiary of such a system

Exclusion Criteria:

1. Significant disease other than COPD. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
2. Clinical relevant abnormal baseline hematology, blood chemistry or urinalysis. If the abnormality defines a disease listed as an exclusion criterion, the patient is excluded
3. Serum glutamic oxaloacetic transaminase (SGOT) >80 IU/L; serum glutamic pyruvic transaminase (SGPT) >80IU/L, bilirubin >2.0mg/dL or creatinine >2.0mg/dL
4. Serum potassium level above or below the normal range
5. Total blood eosinophil count >=600/mm³
6. Recent history (i.e., one year or less) of myocardial infarction
7. Recent history (i.e., three years or less) of heart failure or any cardiac arrhythmia requiring drug therapy
8. History of cancer, other than treated basal cell carcinoma, within the last five years
9. History of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis
10. History of thoracotomy with pulmonary resection. History or a thoracotomy for other reasons should be evaluated as per exclusion criteria no. 1
11. History of asthma, allergic rhinitis or atopy
12. History of or active alcohol or drug abuse
13. Known active tuberculosis
14. Upper respiratory tract infection or COPD exacerbation in the six weeks prior to screening visit or between the screening visit and visit 2
15. Known symptomatic prostatic hypertrophy or bladder neck obstruction
16. Known narrow-angle glaucoma
17. Current significant psychiatric disorders
18. Regular use of daytime oxygen therapy
19. Use of beta-blocker medications, mono-amine oxidase inhibitors or tricyclic antidepressants
20. Use of cromolyn sodium or nedocromil sodium
21. Use of antihistamines.
22. Use of oral corticosteroid medication at unstable doses (i.e., less than six weeks on a stable dose before screening visit or a change between the screening visit and visit2) or at a dose in excess of the equivalent of 10 mg of prednisone per day or 20mg every other day
23. Use of oral beta-adrenergics or long-acting beta-adrenergics such as salmeterol (Serevent®) and formoterol in the two weeks prior to the screening visit or between the screening visit and visit 2
24. Changes in the therapeutic plan within the last six weeks prior to the screening visit or between the screening visit and visit 2, excluding changes from long acting or oral beta-adrenergics to short acting inhaled beta-adrenergics for purposes of this trial
25. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception
26. Known hypersensitivity to anti-cholinergic or beta-agonist drugs or any other component of either Combivent® formulations
27. Use of an investigational drug within one month or six half lives prior to the screening visit
28. Previous participation in this study
29. Patient deprived of their freedom by a judicial or administrative decision
30. Patient leaving in medical or social establishments
31. Patient hospitalized for mental disorder without his (her) consent
32. Patient under guardianship
33. Patient in emergency situations

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2001-04; Primary Completion 2001-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with clinically significant changes in electrocardiogram (ECG) parameters (ventricular rate, PQ, QRS, QT and QTc intervals) | Baseline, up to 8 days after last treatment day
Number of patients with clinically significant changes in vital signs (blood pressure, puls rate, respiratory rate) | Baseline, up to 8 days after last treatment day
Changes in intra ocular pressure (IOP) | Baseline, up to 30 min after last drug administration
Changes in serum potassium levels | Baseline, up to 180 min after last drug administration
Changes in serum glucose levels | Baseline, up to 60 min after last drug administration
Number of patients with clinically significant changes from baseline in clinical laboratory evaluations | Baseline, 8 days after last treatment day
Number of patients with adverse events including paradoxical bronchospasm | Up to 8 days after last treatment day
Number of patients with clinically significant changes from baseline in physical examination | Baseline, 8 days after last treatment day

SECONDARY OUTCOMES:
Change in FEV1 (forced expiratory volume in one second) | Baseline, up to 180 min after last drug administration
Change in FVC (forced vital capacity) | Baseline, up to 180 min after last drug administration